CLINICAL TRIAL: NCT01409395
Title: The Pharmacokinetic Interaction Between Metformin and Nizatidine in Healthy Volunteers
Brief Title: Drug-Drug Interaction Study With Metformin and Nizatidine
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University of California, San Francisco (Other)
Collaborators: National Institute of General Medical Sciences (NIGMS) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 6968; R01GM036780 (NIH)
Record Dates: First submitted 2011-07-29; First posted 2011-08-04 (Estimated); Last update posted 2014-04-10 (Estimated); Status verified 2014-04

CONDITIONS: Healthy
Keywords: Drug drug interaction
MeSH Terms: interventions — Metformin; Nizatidine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Metformin (Experimental): Subjects will be dosed with Metformin alone (850 mg)
  Interventions: Drug: Metformin
- Metformin and Nizatidine (Experimental): Subjects will be dosed with metformin in conjunction with nizatidine
  Interventions: Drug: Metformin and nizatidine

INTERVENTIONS:
Drug: Metformin and nizatidine — Subjects will be given a single oral dose of 850 mg of metformin and a single oral dose of 600 mg of nizatidine
  Other Names: Metformin: Fortamet, Glucophage; Nizatidine: Axid
  Arms: Metformin and Nizatidine
Drug: Metformin — Subjects will be given a single oral dose of 850 mg of metformin
  Other Names: GLUCOPHAGE
  Arms: Metformin

SUMMARY:
This study will address the following question: Does nizatidine affect the pharmacokinetics of metformin in healthy volunteers? Recent studies in the Giacomini laboratory have indicated that nizatidine may block metformin elimination from the kidney by inhibiting organic cation transporter efflux of metformin. The investigators hypothesize that the co-administration of metformin and nizatidine will reduce the renal clearance (CLR) of metformin leading to increased plasma concentrations and potential risk for toxicities. Knowledge of the pharmacokinetic interaction profile of metformin with organic transporter inhibitors, such as nizatidine, is important to help develop safer more effective drug therapy with reduced side effects.

DETAILED DESCRIPTION:
Screening Procedures:

Prior to enrollment, subjects will be asked to come to the Clinical and Translational Science (CTSI) Clinical Research Centre (CRC) at San Francisco General Hospital (SFGH). The study protocol and procedures will be explained in detail, all questions will be answered, and subjects will be provided a consent form to sign. The screening visit will be conducted within 14 days of the first inpatient visit i.e. first metformin alone or metformin with nizatidine dosing day.

Only after subjects have consented to participate in the study will the screening procedures commence. All subjects recruited in this study will have already consented to the pharmacogenomics in ethnically diverse populations (SOPHIE) study, a previously established cohort of healthy people living in San Francisco. A review of the subject's medical history and health questionnaire will be conducted to re-assess health status and confirm eligibility (see attached health questionnaire). Changes in medication or drug use history will be noted during the study.

During the screening visit, vital signs as well as blood and urine samples will be taken from all subjects for laboratory analysis. A single blood sample (10 mL) will be taken by venipuncture to measure a complete blood count (CBC), electrolytes, blood urea nitrogen (BUN), creatinine, and liver function tests (LFTs) to screen for anemia and renal or hepatic insufficiency (see Inclusion/Exclusion Criteria).

Procedures During Main Study:

An equal number of subjects will be randomized, by a computer program, into one of the two study arms described below, prior to their screening visit. After at least a 1-week washout period, subjects will be assigned to the other treatment arm. The duration of the study will consist of two 24-hour inpatient study visits (2 non-consecutive overnight stays), separated by at least 1-week wash out period.

Randomized Study Visit Day 1: Metformin alone Subjects will report to the CRC at approximately 7:30 AM, after an overnight fast of at least 10 hours (fasted from approximately 10:00 PM). Vital signs and a brief history will be taken upon arrival. If all inclusion/exclusion criteria are met, one intravenous (IV) catheter will be inserted into a forearm vein to facilitate blood sampling. An initial blood sample of 10 mL will be drawn (from the IV line) for the determination of plasma metformin, creatinine, and nizatidine concentrations prior to the administration of metformin (i.e. baseline measurement). Next, each subject will receive an oral dose of 850 mg of metformin with 8 oz of water. Blood samples (5 mL each) will then be drawn at 0.5, 1, 1.5, 2, 2.5, 3, 3.5, 4, 6, 8, 10, 12, and 24 hours post-dose for the determination of plasma metformin and nizatidine concentrations. An additional 5 mL of blood will be drawn at the 6-hour and 12-hour time points for the measurement of serum creatinine to allow the calculation of creatinine clearance (CLcr). Blood samples obtained by finger prick will be taken at 0, 0.5, 1, 1.5, 2, 2.5, 3, 3.5 and 4 hours after ingestion of metformin (total of 0.1 mL) to measure blood glucose levels. Additional biomarkers of metformin/nizatidine response and toxicities, such as plasma insulin, glucose and AMPK activation, may also be determined on the blood samples collected. Subjects will remain at the CRC and receive standardized meals starting 4 hours post metformin dosing. Subjects will be discharged and allowed to go home the following morning after the collection of the last (24 hour) blood and urine sample at approximately 8 AM. All blood samples will be centrifuged, and the plasma separated immediately and stored at -80oC until analysis.

Urine collection:Subjects will be asked to void their bladder prior to metformin administration (baseline urine sample) and to drink 8 oz of water every 4 hours to maintain urine flow and pH. Aliquots of urine will be collected for the following time frames: 0-2, 2-4, 4-8, 8-12, and 12-24 hours post metformin dosing. Additionally, aliquots from collections taken between 0-12 and 0-24 hours will be pooled for analysis of creatinine. Subjects will be advised to collect all urine produced during the inpatient visit. The volume and pH of each urine collection will be recorded and an aliquot (20 mL) from each collection period will be stored at -80°C for determination of urinary metformin, creatinine, nizatidine and nizatidine metabolite concentrations.

Randomized Study Visit Day 2:Co-administration of metformin with nizatidine Subjects will report to the CRC after an overnight fast as previously described. After the collection of the baseline blood and urine samples, subjects will receive an oral dose of 600 mg nizatidine and 850 mg of metformin with 8 oz of water. The study procedures described in "Randomized Study Visit Day 1" and "Urine collection" will be repeated.

Study Restrictions:

Concomitant Medications:

The study requires that healthy participants refrain from taking any medications (except for daily vitamins or oral contraceptives) for the duration of the study, in particular medication(s) that interfere with the pharmacokinetics of metformin or nizatidine (See Exclusion criteria 13.7).

Other Study Restrictions:

Subjects will be required to use adequate contraceptive means to avoid pregnancy throughout the study. Subjects must remain within the CRC throughout the two 24 hour inpatient visits unless accompanied by a CRC staff member. Subjects are to refrain from smoking and from ingesting caffeine, alcohol, orange and grapefruit juice containing products from the night before each inpatient study day until the study is complete, approximately 24 hours after dosing.

Clinical and Laboratory Determinations:

Analytical Methods:

Measurement of metformin, creatinine, nizatidine and nizatidine metabolites in plasma and urine will be preformed by High Performance Liquid Chromatography (HPLC) with tandem mass spectrometry (MS/MS), using assays previously described and validated20-22.

Hematology, Blood Chemistry and Urinalysis:

The following standard biochemistry, blood chemistry and urinalysis will be performed at the screening visit:

1. Hematology, (Complete Blood Count with differential, CDP): WBC with differential, red blood cells (RBC), RBC indices (HGB, HCT, MCV, MCH, MCHC) and platelet count.
2. Blood chemistry (Metabolic Comprehensive Panel, METC): sodium, potassium, chloride, carbon dioxide, creatinine, blood urea nitrogen, glucose, calcium, bilirubin (total), phosphate (total), AST, ALT, albumin and alkaline phosphatase
3. Urinalysis: urine protein (dipstick) and blood (dipstick).

Other: Pregnancy test:

A urine test will be administered to females who have had their first menstrual period to make ensure that they are not pregnant. Pregnant females will be excluded from the study.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18-45 years
2. Male or female
3. If female, using appropriate contraception
4. Healthy as judged by medical examination, medical history and normal biochemical and hematological measures
5. Normal urinalysis and renal function
6. Understand the nature and purpose of the study and provide informed consent

Exclusion Criteria:

1. Pregnant or lactating woman (female subjects will have a urine pregnancy test at the screening visit)
2. Abnormal bone marrow function (leukocyte, neutrophil, or platelet counts outside the normal range)
3. History of hypersensitivity or allergic reaction to metformin or nizatidine
4. Risk of congestive heart failure requiring pharmacologic treatment (medical history)
5. History of renal or hepatic dysfunction (e.g., CLcr <60mL/min, ALT >80U/L, AST>60 U/L)
6. Anemic (hemoglobin <12 g/dL)
7. Use of any medications (including over the counter products, herbal products, or mineral supplements) with the exception of a daily vitamin or oral contraceptives. In particular use of medications that are known to interfere with the pharmacokinetics of metformin and nizatidine such as cimetidine, cetirizine, ketoconazole, procainamide, St. John's Wort, and testosterone are prohibited.
8. Laboratory parameters that are more than 2 standard deviations from the laboratory mean
9. Subject carries a MATE2K gene variant that is predicted to effect MATE2K protein expression

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 10 (Actual)
Dates: Start 2011-09; Primary Completion 2013-03 (Actual); Study Completion 2013-03 (Actual)

PRIMARY OUTCOMES:
Composite of Pharmacokinetics of co-administration of nizatidine & metformin in healthy volunteers. | 24 hours
  Cmax and Tmax will be determined from AUC-time curve Glomerular filtration rate (GFR) will be approximated by measured creatinine clearance using the following equation:GFR calculation: GFR = CLcreatinine = (Urinary creatinine * V) / (Plasma creatinine)

CONTACTS AND LOCATIONS:
Overall Officials: Kathleen M Giacomini, Ph.D, Principal Investigator — University of California, San Francisco
Locations (1):
- Ucsf Ctsi Crc, San Francisco, California, United States